CLINICAL TRIAL: NCT01825720
Title: Effect of Glucose-Insulin-Potassium on Hyperlactatemia in Patients Undergoing Valvular Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2012-0347
Record Dates: First submitted 2013-03-26; First posted 2013-04-08 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-10

CONDITIONS: Valvular Heart Disease
Keywords: GIK, valvular heart surgery, lactate
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- (Glucose-Insulin-Potassium)GIK group (Experimental): infusion of 0.1 IU/kg/hr of insulin and mixture of 30% dextrose water with 80 mmol/l of potassium in the rate of 0.5 ml/kg/hr through out the surgery
  Interventions: Drug: (Glucose-Insulin-Potassium)GIK group
- normal saline group (Active Comparator): same rate of normal saline
  Interventions: Drug: normal saline group

INTERVENTIONS:
Drug: (Glucose-Insulin-Potassium)GIK group — infusion of 0.1 IU/kg/hr of insulin and mixture of 30% dextrose water with 80 mmol/l of potassium in the rate of 0.5 ml/kg/hr through out the surgery
  Arms: (Glucose-Insulin-Potassium)GIK group
Drug: normal saline group — same rate of normal saline
  Arms: normal saline group

SUMMARY:
Hyperlactatemia, occuring 10-20% in patients undergoing valvular heart surgery, is known to be associated with hemodynamic instability, organ dysfunction and increased postoperative morbidity and mortality. Glucose-Insulin-Potassium(GIK) has been constantly used as an adjuvant therapy in patients with myocardial infarction or in the patients undergoing valvular heart surgery to reduce the low cardiac output syndrome and mortality. GIK is known to prevent excretion of lactate and to increase the extraction of lactate after reperfusion with various mechanism. In addition, it is also known to decrease ischemic-reperfusion injury of myocardium after CPB, to improve myocardial contractility, insulin resistance and hyperglucemia. As a result, it brings hemodynamic stability and sufficient oxygen supply to the tissue, which might reduce the incidence of hyperlactatemia after valvular heart surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients(20 yr or older) undergoing elective valvular heart surgery under cardiopulmonary bypass(CPB) with more than 2 of following features:

  1. congestive heart failure
  2. infective endocarditis
  3. redo valvular surgery
  4. surgery combined with coronary bypass graft
  5. multiple valvular surgery
  6. expected CPB duration longer than 2 hr 7> preoperative serum creatinine over 1.4 mg/dl 8> preoperative hemoglobin level less than 12 mg/dl 9> left ventricular ejection fraction less than 40%

Exclusion Criteria:

1. emergency surgery
2. hemodynamic instability before surgery (mean arterial pressure < 60 mmHg, heart rate >100 /min
3. need for pharmacological or mechanical assist for hemodynamic stability before surgery
4. baseline blood lactate level more than 2 mmol/l
5. on steroid or NSAID
6. hepatic dysfunction

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2013-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
perioperative blood lactate level | change of blood lactate level for 10 time points (before induction of anesthesia, immediately after induction of anesthesia, pre-CPB, 15 min after CPB, ACC off, post-CPB, sternum closure, ICU admission, 3 h after ICU admission, POD 1)
  Measuring blood lactate level at each time point to compare the efficacy of GIK solution between control and Gik group

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Roh GU, Shim JK, Song JW, Kang HM, Kwak YL. Effect of glucose-insulin-potassium on hyperlactataemia in patients undergoing valvular heart surgery: A randomised controlled study. Eur J Anaesthesiol. 2015 Aug;32(8):555-62. doi: 10.1097/EJA.0000000000000250. PMID 25760680